CLINICAL TRIAL: NCT04373616
Title: A Phase 2 Double-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability and Target Engagement of ACI-24 in Adults With Down Syndrome
Brief Title: A Study of ACI-24 in Adults With Down Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: decision to proceed with an optimized study design and optimized vaccine formulation
Sponsor: AC Immune SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACI-24-DS-1902; 2020-000634-18 (EudraCT Number)
Record Dates: First submitted 2020-04-27; First posted 2020-05-04 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Down Syndrome
Keywords: Alzheimer related disease; Cognitive decline
MeSH Terms: conditions — Down Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACI-24 (Experimental)
  Interventions: Biological: ACI-24
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ACI-24 — injections
  Arms: ACI-24
Biological: Placebo — injections
  Arms: Placebo

SUMMARY:
This study is a prospective multicenter, placebo-controlled, double-blind, randomized study to assess the effect of one dose ACI-24 versus placebo over a 74-week treatment period and 26-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with DS with a cytogenetic diagnosis being either trisomy 21 or complete unbalanced translocation of the chromosome 21.
2. Age ≥ 40 and ≤ 50 years at screening.
3. Elevated brain Aβ as evidenced by composite SUVR ≥ 1.25 on florbetaben PET scan assessed by central reading.
4. Subjects, their legal representatives (if applicable) and/or their study partners in the opinion of the investigator, are able to understand and to provide written informed consent before starting any study-related activities.
5. In the opinion of the investigator, subjects, their legal representatives (if applicable) and/or their study partners are able to fully participate in the study, be sufficiently proficient in the official languages(s) of the country they are living in, and be capable of reliably completing study assessments.
6. Mild to moderate intellectual disability as per Diagnostic and Statistical Manual of Mental Disorders (DSM-5) classification.
7. Subjects must have a study partner who has direct and regular contact with the subject and who is able to provide reliable answers to questions related to the subject, according to the study investigator.
8. Subjects in preclinical stage of AD or with mild cognitive impairment due to AD.

Exclusion Criteria:

1. Clinical diagnosis of AD dementia in DS as per International Classification of Diseases 10 (ICD-10).
2. DSQIID > 20.
3. Intelligence quotient score ≤ 40 (KBIT-2).
4. Diagnosis of autism spectrum disorder or any other unstable/uncontrolled psychiatric or neurologic illness other than DS.
5. Any unstable and/or clinically significant medical condition likely to hamper the evaluation of safety and/or efficacy of the study vaccine (eg, severe and untreated obstructive sleep apnea, clinically significant reduction in serum B12 or folate levels, clinically significant abnormalities of thyroid function, stroke or other cerebrovascular conditions), as per investigator's judgement.
6. Subjects considered to be unable to complete any study exams and assessments (eg, because of significant hearing or visual impairments or other disabilities), according to the investigator, and potentially affecting study compliance.
7. DSM-5 criteria for drug or alcohol abuse or dependence currently met within the past 5 years.
8. History or presence of uncontrolled seizures. If history of seizures, they must be well controlled with no occurrence of seizures in the 2 years before study screening. The use of antiepileptic medications is permitted.
9. History of meningitis or meningoencephalitis.
10. History of moderate or severe traumatic brain injury.
11. History of cancer within the past 5 years other than treated squamous cell carcinoma, basal cell carcinoma and melanoma in-situ, in-situ prostate cancer, or in-situ breast cancer which have been fully removed and are considered cured.
12. History of inflammatory neurological disorders.
13. History of autoimmune disease with potential for central nervous system involvement.
14. Severe infections or a major surgical operation within 3 months before screening.
15. History of chronic or recurrent infections judged to be clinically significant by the investigator and would potentially hamper the evaluation of efficacy and safety assessments.
16. History or presence of immunological or inflammatory conditions judged to be clinically significant by the investigator.
17. History of severe allergic reaction (eg, anaphylaxis) including, but not limited to, severe allergic reaction to previous vaccines, foods, and/or medications.
18. Clinically significant abnormal vital signs including sustained sitting blood pressure greater than 160/90 mm Hg.
19. Subjects who have donated blood or blood products in the 30 days before screening or who plan to donate blood while participating in the study or within 4 weeks after completion of the study.
20. Subjects with diabetes mellitus with hemoglobin A1c (HbA1c) levels of ≥ 8.0%.
21. Any contraindication for lumbar puncture for those subjects consenting to the optional lumbar puncture.
22. MRI scan at screening showing a single area of cerebral vasogenic edema, superficial siderosis, or evidence of a previous macrohemorrhage or showing more than 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"). Evidence of space-occupying lesions other than benign meningioma of less than 1 cm diameter, more than 2 lacunar infarcts, or 1 single infarct larger than 1 cm in diameter. Screening MRI scan showing structural evidence of alternative pathology not consistent with AD and is considered to be at the origin of subject's symptoms.
23. In the opinion of the site investigator, deviations from normal values for hematologic parameters, liver function tests, and other biochemical measures, judged to be clinically significant by the investigator.
24. Subjects with a positive Human Immunodeficiency Virus (HIV) test at screening.
25. Subjects with clinical or laboratory evidence of active Hepatitis B or C at screening.
26. Subjects with positive syphilis serology consistent with active syphilis at screening.
27. Clinically significant arrhythmias or other abnormalities on ECG at screening (minor abnormalities documented as clinically insignificant by the investigator are allowed).
28. Any vaccine received within the 2 weeks before screening, including influenza vaccine.
29. Subjects with treated hypothyroidism not on a stable dose of replacement medication for at least 3 months before screening and having clinically significant abnormal serum T4 and/or thyroid-stimulating hormone at screening.
30. Subjects who have been receiving any experimental drug with a washout less than 30 days or less than 5 half-lives of the drug, whichever is longer.
31. Subjects being treated with any anticoagulants or antiplatelet drugs, except aspirin at doses of 100 mg daily or lower.
32. Use of antidepressants (other than selective serotonin reuptake inhibitors/serotonin-norepinephrine reuptake inhibitors at stable dose); antipsychotics (typical or atypical); γ-aminobutyric acid agonists (eg, gabapentin); or stimulants (eg, methylphenidate, modafinil). Stable doses of atypical antipsychotics or benzodiazepines are only allowed if this is not considered to influence the assessments, the safety, and the efficacy of the study vaccine according to the site investigator and the site monitor.
33. Current use of anticholinergic agents for bladder dysfunction (eg, oxybutynin, tolterodine, darifenacin, solifenacin, trospium, or fesoterodine) or subjects who have received such treatments within a time period corresponding to 5 half-lives of the respective agent before screening.
34. Chronic use of opioid analgesics. However, limited treatment duration for acute conditions until 24 hours before cognitive assessment is allowed.
35. Current use of antihistaminic agents, especially of first generation. Limited use of second-generation antihistaminics for acute conditions is allowed if not anticipated to influence the cognitive assessments, according to the investigator.
36. Current use of immunosuppressant or immunomodulating drugs or their use within the 6 months before study screening. Current use of oral steroids or their use within the 3 months before study screening.
37. Previous treatment with ACI-24 or any other passive or active immunotherapy against AD and/or for neurological disorders (passive immunization within the 6 months before screening, active immunization at any time point) unless there is firm evidence that the subject was treated with placebo only, and the placebo formulation is not expected to induce any specific immune response.
38. Use of acetylcholinesterase inhibitors or use of glutamatergic drugs (eg, memantine, topiramate, lamotrigine) if not on stable dose for at least 2 months before screening.
39. Concomitant participation in any other clinical study using an investigational drug.
40. Female subjects who are pregnant as confirmed by serum testing at screening or who are planning to become pregnant or lactating.
41. Female or male subjects not using a reliable method of contraception during the treatment period and for 26 weeks (6 months) after the last administration of study vaccine.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) assessed by intensity (mild, moderate or severe) and causal relationship (unrelated, unlikely, possibly or probably related). | from screening up to week 100
Mean change from baseline in systolic and diastolic blood pressure (mmHg) | from baseline up to week 100
Mean change from baseline in heart rate (bpm) | from baseline up to week 100
Mean change from baseline in body temperature (degree Celsius) | from baseline up to week 100
Number of participants reporting suicidal ideation or behavior using Columbia-Suicide Severity Rating Scale (C-SSRS) | from baseline up to week 100
Number of participants with abnormal MRI results | from baseline up to week 100
  Occurrence of Amyloid-related imaging abnormalities (ARIA)

SECONDARY OUTCOMES:
Change from baseline of composite standardized uptake value ratio (SUVR) assessed by amyloid PET imaging using florbetaben | from baseline up to week 76
Change from baseline in anti-Aβ antibody titers in blood | from baseline up to week 100
Change from baseline of amyloid-related biomarkers (Aβ1-40, Aβ1-42), total tau, phosphorylated tau and NfL in blood/CSF (in pg/ml) (CSF is optional) | from baseline up to week 100
Change from baseline of brain tau load assessed by tau PET imaging | from screening up to week 74
Change from baseline of cognitive performance using Cambridge Neuropsychological Test Automated Battery - Paired Associates Learning [CANTAB-PAL] | from baseline up to week 100
  Score is a z-score ranging from -7.5 to 0. A higher score (eg., 0) indicates a better outcome.
Change from baseline of cognitive performance using Cambridge Cognitive Examination - Down Syndrome [CAMCOG-DS] | from baseline up to week 100
  The total score ranges from 0 to 107. A higher score indicates a better outcome.
Change from baseline in adaptive behavior (Vineland Adaptive Behavior Scale) | from baseline up to week 100
  The composite score ranges from 20 to 140. A higher score indicates a better outcome.
Change from baseline in Clinical Global Impression of Change (CGIC) | from baseline up to week 100
  The score ranges from 1 to 7. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Rafii, MD, PhD, Principal Investigator — Alzheimer's Therapeutic Research Institute USC Keck School of Medicine of the University of Southern California, San Diego, CA, USA

IPD SHARING:
Plan to Share IPD: Undecided